CLINICAL TRIAL: NCT05412355
Title: Effects of Incomplete Enhanced Recovery After Surgery Program on Long-term Survival of Patients Undergoing Colorectal Cancer Surgery
Brief Title: Effects of Incomplete ERAS on Clinical Outcomes in Patients With Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xiaogang Shu, Prof., Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: UHCT22040
Record Dates: First submitted 2022-06-06; First posted 2022-06-09 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Colorectal Neoplasms; Enhanced Recovery After Surgery
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Incomplete ERAS: Incomplete ERAS was defined as ERAS compliance < 70%.
  Interventions: Procedure: ERAS protocol
- Non-ERAS: non-ERAS was defined as not executing any ERAS programs.
  Interventions: Procedure: ERAS protocol

INTERVENTIONS:
Procedure: ERAS protocol — ERAS protocol is a series of procedures that enhance the recovery of surgical patients. Patients were grouped according to whether the procedure was attempted.

SUMMARY:
Enhanced recovery after surgery (ERAS) has been reported to be associated with improved outcomes in many studies, most of which involve short-term effects. Only a few studies have reported the long-term effects of highly compliant ERAS. However, to the best of our knowledge, there are no large-scale comparisons between incomplete ERAS (compliance < 70%) and non-ERAS. The aim of this comparative study is to analyze and evaluate the long-term outcomes of incomplete ERAS in laparoscopic colorectal cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* 1. age older than 18 years;2. pathological diagnosis of colorectal cancer;3. radical surgery was performed; and 4. laparoscopic surgery was performed.

Exclusion Criteria:

* 1. ERAS compliance ≥70%; 2. open surgery; 3. switch to laparotomy after laparoscopic surgery; 4. pregnancy or lactation; 5. severe mental illness; 6. Simultaneous malignant tumors of multiple organs; 7. History of other malignant tumors; and 8. Emergency radical colorectal resection due to obstruction, perforation or bleeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this study, we are going to collect clinical data of patients undergoing laparoscopic radical surgery from four large hospitals between August 2008 and December 2016.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-08-10 (Estimated); Study Completion 2022-10-10 (Estimated)

PRIMARY OUTCOMES:
long-term survival | Each patient will be followed for 5 years or until death
  5-year Disease free survival and overall survival

SECONDARY OUTCOMES:
Postoperative complications | within 30 days after surgery
  Postoperative complications within 30 days after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaogang Shu, MD.，PHD., Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (2):
- China (2):
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology., Wuhan, Hubei
  - Union Hospital，Tongji Medical College, Huazhong University of Science and Technology., Wuhan, Hubei

IPD SHARING:
Plan to Share IPD: Yes
After the funders finished the study,the data will be available，if approved by PI.
Supporting Information: Study Protocol
Time Frame: After 2025.1.1
Access Criteria: Approved by PI